CLINICAL TRIAL: NCT02723474
Title: A Single-Centre Pilot Study Exploring the Utility of Magnetic Resonance Imaging in Patients With Chronic Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: ROB0010
Record Dates: First submitted 2015-12-07; First posted 2016-03-30 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2024-06

CONDITIONS: Lung Disease
Keywords: Magnetic Resonance Imaging; Pulmonary Function
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI at baseline and over time (Other): Patients with chronic lung disease will undergo pulmonary function tests, hyperpolarized Helium and or Xenon MRI at each visit.
  Interventions: Device: MRI at baseline and over time

INTERVENTIONS:
Device: MRI at baseline and over time — Hyperpolarized noble gas MRI has been used to explore structural and functional relationships in the lung in patients with lung disease and healthy controls. In contrast to proton-based MRI, Helium-3 and Xenon-129 gas is used as a contrast agent to directly visualize ventilation. Whereas the normal density of gas is too low to produce an easily detectable signal, this is overcome by artificially increasing the amount of polarization per unit volume using optical pumping.

SUMMARY:
Male and female subjects age 18-85 with lung disease will inhale 5ml/kg (patient body weight) hyperpolarized helium and will be scanned using MRI at 3 Tesla, to evaluate the Apparent Diffusion Coefficient (ADC), ventilation defect volume and percent ventilation.

DETAILED DESCRIPTION:
Briefly, during a one to two hour visit, subjects will provide written informed consent and then undergo:

1. brief medical history and vital signs,
2. full pulmonary function tests,
3. proton MRI,
4. spin-density and/or diffusion weighted Helium-3 MRI.

Full pulmonary function tests including spirometry, plethysmography and diffusing capacity of carbon monoxide (DLCO), Lung Clearance Index (LCI) and Airwave Oscillometry (AO) will be performed according to ATS guidelines. MedGraphics Elite Series, MedGraphics Corporation. St. Paul, MN USA and/or nDD EasyOne Spirometer, nDD Medical Technologies Inc. Andover, MA USA will be used. All measurements will be performed in the Pulmonary Function Laboratory at Robarts Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 18-75 with diagnosed lung disease including but not limited to: asthma, emphysema, Chronic Obstructive Pulmonary Disease (COPD), bronchiectasis, sarcoidosis, pulmonary fibrosis, alpha 1-anti-trypsin deficiency, lymphangioleiomyomatosis (LAM) and Bronchiolitis obliterans organizing pneumonia (BOOP)
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject must be able to perform a breathhold for 16s.
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have Forced Expiratory Volume in one second (FEV1) values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater.)
* FEV1 >25% predicted
* Forced Vital Capacity (FVC) > 25% predicted and >0.5Liters

Exclusion Criteria:

* Subject with a contraindication to Magnetic Resonance Imaging (i.e. ferrous implants, cardiac pacemakers). This will be determined through a screening form.
* Subject has a daytime room air oxygen saturation <90% while lying supine.
* Subject unable to tolerate MRI due to patient size and/or known history of claustrophobia.
* Subject previously injured by a metallic object that was not removed.
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Lung function as measured using inhaled gas MRI ventilation defect percent (VDP) | 5 years
  Lung function will be measured using inhaled gas MRI ventilation defect percent

SECONDARY OUTCOMES:
Lung microstructure as measured using inhaled gas MRI Apparent Diffusion Coefficients (ADC) | 5 years
  Lung microstructure as measured using inhaled gas MRI ADC

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Westcott A, Capaldi DPI, McCormack DG, Ward AD, Fenster A, Parraga G. Chronic Obstructive Pulmonary Disease: Thoracic CT Texture Analysis and Machine Learning to Predict Pulmonary Ventilation. Radiology. 2019 Dec;293(3):676-684. doi: 10.1148/radiol.2019190450. Epub 2019 Oct 22. PMID 31638491
- [Derived] Kirby M, Eddy RL, Pike D, Svenningsen S, Coxson HO, Sin DD, McCormack DG, Parraga G; Canadian Respiratory Research Network. MRI ventilation abnormalities predict quality-of-life and lung function changes in mild-to-moderate COPD: longitudinal TINCan study. Thorax. 2017 May;72(5):475-477. doi: 10.1136/thoraxjnl-2016-209770. Epub 2017 Mar 3. PMID 28258250